CLINICAL TRIAL: NCT06054815
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel, Phase 2a Clinical Trial to Evaluate the Efficacy and Safety of DA-1241 in Subjects With Presumed Non-alcoholic Steatohepatitis (NASH)
Brief Title: Study to Evaluate the Efficacy and Safety of DA-1241 in Subjects With Presumed NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA1241_NASH_IIa
Record Dates: First submitted 2023-09-05; First posted 2023-09-26 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: NON-ALCOHOLIC STEATOHEPATITIS
Keywords: NASH; NON-ALCOHOLIC STEATOHEPATITIS
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — DA-1241; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 Group 1 (Experimental): DA-1241 Dose 1
  In Part 1: Participants will be randomized into 3 treatment groups and will be dosed with: DA-1241 or placebo in a 1:2:1 ratio.
  Interventions: Drug: DA-1241; Drug: DA-1241 Placebo; Drug: Sitagliptin Placebo
- Part 1 Group 2 (Experimental): DA-1241 Dose 2
  In Part 1: Participants will be randomized into 3 treatment groups and will be dosed with: DA-1241 or placebo in a 1:2:1 ratio.
  Interventions: Drug: DA-1241; Drug: Sitagliptin Placebo
- Part 1 Group 3.1 (Placebo Comparator): DA-1241 Placebo and Sitagliptin Placebo
  In Part 1: Participants will be randomized into 3 treatment groups and will be dosed with: DA-1241 or placebo in a 1:2:1 ratio.
  Interventions: Drug: DA-1241 Placebo; Drug: Sitagliptin Placebo
- Part 2 Group 3.2 (Placebo Comparator): DA-1241 Placebo and Sitagliptin Placebo
  In Part 2: Participants will be randomized into 2 treatment groups and will be dosed with: DA-1241 in combination with sitagliptin (DA-1241/sitagliptin) or DA-1241/ sitagliptin placebo in a 2:1 ratio.
  Interventions: Drug: DA-1241 Placebo; Drug: Sitagliptin Placebo
- Part 2 Group 4 (Experimental): DA-1241 and Sitagliptin
  In Part 2: Participants will be randomized into 2 treatment groups and will be dosed with: DA-1241 in combination with sitagliptin (DA-1241/sitagliptin) or DA-1241/ sitagliptin placebo in a 2:1 ratio.
  Interventions: Drug: DA-1241; Drug: Sitagliptin

INTERVENTIONS:
Drug: DA-1241 — Route of Administration: Oral, with subjects in a fasting state
  Arms: Part 1 Group 1; Part 1 Group 2; Part 2 Group 4
Drug: Sitagliptin — Route of Administration: Oral, with subjects in a fasting state
  Arms: Part 2 Group 4
Drug: DA-1241 Placebo — Route of Administration: Oral, with subjects in a fasting state
  Arms: Part 1 Group 1; Part 1 Group 3.1; Part 2 Group 3.2
Drug: Sitagliptin Placebo — Route of Administration: Oral, with subjects in a fasting state
  Arms: Part 1 Group 1; Part 1 Group 2; Part 1 Group 3.1; Part 2 Group 3.2

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, parallel, Phase 2a clinical trial to evaluate the efficacy and safety of DA 1241 in subjects with presumed non-alcoholic steatohepatitis (NASH).

DETAILED DESCRIPTION:
Clinical trial DA1241_NASH_IIa is a multicenter, randomized, double-blind, placebo-controlled, parallel-arm, Phase 2a clinical trial to evaluate the efficacy and safety of DA-1241 in subjects with presumed NAFLD.

Part 1 of this clinical trial intends to explore the efficacy of DA-1241 in subjects with NASH after administration of oral DA-1241 at varying doses or identical placebo in 3 treatment groups for 16 weeks/112 days.

Part 2 intends to explore the efficacy of DA-1241 in subjects with NASH after administration of oral DA-1241 in combination with sitagliptin versus an identical placebo for 16 weeks/112 days.

ELIGIBILITY:
Inclusion Criteria

1. Subjects who are able to understand and sign informed consent before the conduct of any protocol specific screening procedures.
2. Subjects who are male or female, aged 18 to 75 years inclusive at the time of consent.
3. Female subjects of childbearing potential:

   1. Must agree to abide by contraception requirements, must not be lactating, and avoid pregnancy during study participation from the first Screening visit until 30 days after the last dose of study drug.
   2. Must commit to an additional method of birth control in addition to male partners agreeing to use condoms with spermicide, throughout the study including for at least 30 days after the last dose of the study drug:

      * True abstinence: Refraining from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [eg, calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable).
      * Combined (containing estrogen and progestogen) hormonal birth control (oral, intravaginal, injectable, or transdermal) associated with inhibition of ovulation initiated at least 30 days before dose administration.
      * Progestogen only hormonal birth control (oral, injectable, or implantable) associated with inhibition of ovulation initiated at least 30 days before study dose administration.
      * Bilateral tubal occlusion/ligation.
      * Intrauterine device (IUD).
      * Intrauterine hormone releasing system (IUS).
      * Vasectomized partner.
4. Female subjects of non-childbearing potential do not need to use birth control during or after study drug treatment if considered of non-childbearing potential due to any of the following criteria:

   1. Premenopausal female with permanent sterility or permanent infertility as due to one of the following:

      * Permanent sterility due to a hysterectomy, bilateral salpingectomy, bilateral oophorectomy.
      * Non-surgical permanent infertility due to Mullerian agenesis, androgen insensitivity, or gonadal dysgenesis; Investigator discretion should be applied to determining study entry for these individuals.
   2. Postmenopausal female subjects, with no menses for 12 or more months without an alternative medical cause AND a follicle stimulating hormone (FSH) level ≥ 40 IU/L.
5. Male subjects who are sexually active with a female partner of childbearing potential must agree to use male condoms and spermicide, even if the male subject has undergone a successful vasectomy (males with vasectomy can use condoms without spermicide), from Day 1 until at least 30 days after the last dose of the study drug.
6. Subjects with a BMI > 23 kg/m2 at first Screening Period visit.
7. Subjects with a qualifying ALT result (40 IU/L ≤ ALT < 200 IU/L) as determined by the laboratory assessment at the first Screening Period visit.
8. Subjects with a confirmed NASH diagnosis or conditions consistent with NASH.
9. Subjects with an HbA1c ≥ 5.7% and < 9.5% (5.7% ≤ HbA1c < 9.5%).
10. Subjects with ≥ 8% hepatic fat on MRI after confirming a qualifying ALT result at Screening.
11. Subjects with CAP score by FibroScan® of ≥ 290 dB/m at the time of the first Screening Period visit.
12. Subjects with 7 kPa ≤ VCTE score by FibroScan® < 14 kPa at the time of the first Screening Period visit.
13. For subjects receiving stable doses of the following medications prior to the first Screening Period visit, the following conditions applied:

    1. Sodium-glucose cotransporter-2 (SGLT-2): no dose changes for at least 12 weeks prior to the first Screening Period visit.
    2. Insulin and oral antidiabetic medications or drugs for dyslipidemia: no dose changes for at least 8 weeks prior to the first Screening Period visit; defined as a change of no more than a ± 25% in total daily dose of insulin during this period.
    3. Vitamin E > 400 I/U: daily dose of ≤ 800 I/U, stable for at least 12 weeks prior to the first Screening Period visit.
    4. HMG-CoA Reductase Inhibitor (statins): no dose changes for at least 8 weeks prior to the first Screening Period visit.

Exclusion Criteria

1. Subjects who have used an investigational agent within 30 days or 5 elimination half-lives; whichever is longer prior to the first Screening Period visit.
2. Subjects diagnosed with liver disease other than NASH (eg, chronic viral hepatitis, decompensated cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, α-1-antitrypsin deficiency, primary biliary cholangitis, drug-induced liver disease).
3. Subjects who have a positive test result for hepatitis A virus immunoglobulin M, hepatitis B surface antigen, hepatitis B core antibody, hepatitis C virus antibody, or reactive human immunodeficiency virus (HIV) after providing a qualifying ALT result at the first Screening Period visit, or who have a known history of HIV infection. However, subjects with a positive hepatitis C virus antibody could be eligible after undergoing reflex testing (HCV-RNA negative) and evaluation by the Investigator.
4. Clinically significant laboratory results as evaluated by the Investigator after providing a qualifying ALT result at the first Screening Period visit. Subjects will be excluded if:

   1. AST ≥ 200 U/L
   2. Platelets ≤ 150,000/mm3
   3. Albumin < 3.8 g/dL
   4. Total bilirubin ≥ 1.5 mg/dl, except with clinical diagnosis of Gilbert's syndrome
   5. Direct bilirubin > 0.3 mg/dL
   6. Phosphatidylethanol > 40 ng/mL
   7. INR > 1.3 in the absence of anticoagulants
5. Subjects with an estimated glomerular filtration rate < 60 mL/min/1.73m2 based on modification of Diet in Renal Disease (MDRD) formula.
6. Subjects with a corrected QT interval by Fridericia (QTcF) of > 450 ms in males, and > 470 ms in females.
7. Subjects who are taking one or more of the following medications:

   1. Within 12 weeks prior to the first Screening Period visit: i. Medication that is known to cause or worsen fatty liver disease (amiodarone, valproate, tamoxifen, methotrexate, etc.) for > 14 days. ii. Medication for weight loss. iii. Chronic use of systemic corticosteroids for > 14 days; however, administration of intranasal, topical, or inhaled corticosteroids is allowed. iv. DPP-4 inhibitors, thiazolidinediones (TZDs), or GLP-1 agonists.
   2. St. John's Wort or consuming grapefruit juice within 2 weeks prior to the first Screening Period visit.
   3. Digoxin, strong CYP3A4 inhibitors (a ≥ 10-fold increase in AUC of sensitive substrate), or strong CYP3A4 inducers (decreases the AUC of sensitive index substrates of a given metabolic pathway ≥ 80% increase) received within 5 half-lives or 14 days (whichever is longer) prior to the first Screening Period visit.
8. Subjects who cannot get an MRI scan.
9. Subjects who have a history of cirrhosis, a VCTE ≥ 14 kPa, portal hypertension as evidenced by a history of splenomegaly > 15 cm, ascites, hepatic encephalopathy, varices on imaging/endoscopy or history of variceal bleeding, or a Model for End Stage Liver Disease (MELD) score > 10.
10. Subjects who have undergone bariatric surgery within 5 years prior to the first Screening Period visit after confirming a qualifying ALT result or are planning bariatric surgery during the clinical trial.
11. Subjects with a history of malignancy within 2 years prior to the first Screening Period visit. However, subjects who have completed all cancer therapies with no evidence of active malignancy within the 2 years prior to the first Screening Period visit will be allowed, except for squamous cell or basal cell carcinoma of the skin definitively treated > 12 weeks prior to the first Screening Period visit.
12. Subjects who have a presence of clinically significant cardiac (including Grade III/IV heart failure as defined by the New York Heart Association Criteria [Appendix 10.2]). This includes subjects with a history of myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass graft, or stroke within 90 days prior to the first Screening Period visit.
13. Subjects with a history of acute cardiovascular disease (uncontrolled arrhythmia, unstable angina, myocardial infarction, stroke, transient ischemic attack, cerebrovascular disease, etc.) within 12 weeks prior to the first Screening Period visit.
14. Subjects with a history of drug abuse or alcohol addiction within 12 weeks prior to the first Screening Period visit.
15. Subjects with a positive screen for drugs of abuse (ie, amphetamines, barbiturates, benzodiazepines, cocaine, methadone, opiate metabolite, and phencyclidine). Subjects who have been prescribed benzodiazepine or opiates for stable chronic medical illness may still qualify for the study at the discretion of the Investigator and review of the Medical Monitor.
16. Subjects who have physical (severe disorders in liver, heart, kidney, lung, blood, endocrine system, musculoskeletal system, gastrointestinal system, etc.) or mental (cognitive impairment, mental illness) conditions that may affect the subject's ability to participate in the clinical trial.
17. If female, subjects who are pregnant or lactating or intend to become pregnant during the clinical trial.
18. If male, subjects who intend to impregnate a partner.
19. Subjects who intend to donate ova or sperm during the clinical trial.
20. Subjects with known or suspected intolerance or hypersensitivity to IPs, closely-related compounds, or any of the stated ingredients.
21. Subjects with a weight change of > 10% measured at the first Screening Period and TP1 visits.
22. Subjects who cannot communicate reliably with the Investigator or are unlikely to cooperate with the requirements of the clinical trial.
23. Subjects with any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject's participation in, or completion of, the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change alanine transaminase (ALT) levels | Baseline to Day 112
  To explore the efficacy (change from baseline in alanine transaminase [ALT]) of DA-1241 in subjects at risk of NASH or subjects with non-alcoholic fatty liver disease (NAFLD) after administration of oral DA-1241 at varying doses of placebo and in combination with sitagliptin.

SECONDARY OUTCOMES:
ALT Normalization | Baseline to Day 112
  Proportion of subjects with normalization of ALT: < 30 IU/L
AST, GGT, ALP | Baseline to Day 112
  Absolute change in aspartate transaminase (AST), gamma glutamyl transpeptidase (GGT), and alkaline phosphatase (ALP).
Total cholesterol, LDL, HDL, triglyceride, and free fatty acids | Baseline to Day 112
  Absolute change in total cholesterol, low and high-density lipoprotein cholesterol, triglyceride, and free fatty acids from baseline.
A1c | Baseline to Day 112
  Absolute change in hemoglobin A1c (HbA1c) (%).
Glucose | Baseline to Day 112
  Absolute change in fasting plasma glucose (mg/dL).
Fasting insulin | Baseline to Day 112
  Absolute change in fasting insulin.
HOMA-IR | Baseline to Day 112
  Absolute change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR).
Adipo-IR | Baseline to Day 112
  Absolute change in adipose tissue insulin resistance index (adipo-IR).
CAP | Baseline to Day 112
  Absolute change in controlled attenuation parameter (CAP) score assessed by FibroScan®.
VCTE | Baseline to Day 112
  Absolute change in vibration-controlled transient elastography (VCTE) score assessed by FibroScan®.
FAST | Baseline to Day 112
  Absolute change in FibroScan®- AST (FAST) score.
Body weight | Baseline to Day 112
  Absolute change in body weight.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Southern California Research Center, Coronado, California
  - Catalina Research Institute, LLC, Montclair, California
  - Velocity Clinical Research, Panorama City, Panorama City, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Integrity Clinical Research, LLC, Doral, Florida
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - GI Associates & Endoscopy Center, Flowood, Mississippi
  - AIG Digestive Disease Research, Florham Park, New Jersey
  - South Texas Research Institute - A Pinnacle Entity, Edinburg, Texas
  - Dallas Research Institute, LLC, Farmers Branch, Texas
  - Pinnacle Clinical Research - Georgetown, Georgetown, Texas
  - Pioneer Research Solutions Inc., Houston, Texas
  - American Research Corporation, San Antonio, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas
  - Apex Mobile Clinical Research, LLC, San Antonio, Texas
  - Liver Institute Northwest, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No